CLINICAL TRIAL: NCT03819283
Title: Prevalence and Impact of NAFLD in Patients With Symptomatic Coronary Artery Disease
Brief Title: NASH and Coronary Disease
Acronym: CORO-NASH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institute of Cardiometabolism and Nutrition, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP180013; 2018-A01752-53 (Other: ANSM)
Record Dates: First submitted 2019-01-10; First posted 2019-01-28 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-03

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: fatty liver, coronary artery disease, atherosclerosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Coronary Artery Disease; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hepatic evaluation (Other)
  Interventions: Diagnostic Test: Hepatic evaluation

INTERVENTIONS:
Diagnostic Test: Hepatic evaluation — Evaluation of hepatic steatosis and fibrosis by non invasive tests, either serum markers (steatotest, Fibrotest) or imaging methods (CAP, FibroScan)

SUMMARY:
Although the clinical relationship between NAFLD/NASH and cardiovascular (CV) risk is now well established, there is very little awareness of the hepatic disease and the way it may contribute to increased CV risk in patients seen in cardiology clinics for complications of coronary artery disease. Our clinical hypothesis is that NAFLD, possibly at a stage of advanced fibrosis, is common in patients with symptomatic coronary artery disease (CAD) and increases the risk of severe atherosclerotic lesions. The primary aim of this study is to determine (a) the prevalence and (b) the severity spectrum of NAFLD among patients with symptomatic coronary artery disease. The secondary aims are: to analyze the impact of the presence and the severity spectrum of NAFLD (steatosis, steatohepatitis and fibrosis) on the severity of CAD ; To determine the profile of NAFLD patients at risk to develop coronary lesions; To explore the mechanistic link between NAFLD and CAD beyond common metabolic risk factors.

DETAILED DESCRIPTION:
Because of shared metabolic risk factors and pathogenic pathways (insulin resistance, chronic low grade inflammation, atherogenic dyslipidemia) non-alcoholic fatty liver disease is frequently associated with cardiovascular (CV) disease. Despite a lot of transversal studies showing a frequent association between NAFLD and CV disease, it is difficult to determine if NAFLD plays an active role in atherogenesis or is just a marker of common risk factors. Some longitudinal studies, although retrospectives, showed that NAFLD favors the progression of early atherosclerosis, suggesting that NAFLD is an independent CV risk factor beyond the association driven by metabolic syndrome.

Although the clinical relationship between NAFLD/NASH and CV risk is now well established, there is very little awareness of the hepatic disease and the way it may contribute to increased CV risk in patients seen in cardiology clinics for complications of coronary artery disease (CAD). Our clinical hypothesis is that NAFLD, possibly at a stage of advanced fibrosis, is common in patients with symptomatic CAD and increases the risk of severe atherosclerotic lesions.

The primary aim of this study is to determine (a) the prevalence of NAFLD among patients with symptomatic CAD.

The secondary aims are:

* To determine the severity spectrum of NAFLD among patients with coronary artery disease.
* To analyze the impact of the presence and the severity spectrum of NAFLD (steatosis, steatohepatitis and fibrosis) on the severity of CAD and long term clinical outcomes (ancillary studies)
* To determine the clinical profile of NAFLD patients at risk to develop coronary lesions
* To explore the mechanistic link between NAFLD and CAD beyond common metabolic risk factors.
* Establish a cohort of patients with NAFLD and coronary disease allowing future subsequent ancillary studies.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old) that undergo coronary angiography for suspected CAD for: acute coronary syndrome (ACS) with ST-elevation ACS (STE-ACS) or non-ST elevation (NSTE-ACS) with or without troponin elevation OR suspicion of stable coronary artery disease after stress imaging techniques and/or symptoms of angina.
* Patients with one or more of traditional cardiovascular risk factors.

Exclusion Criteria:

* Patients unable to sign the informed consent
* Morbidly obese patients (BMI > 40kg/m2)
* Excessive alcohol consumption of more than 50 g/day
* Patients with known other causes of chronic liver disease (viral hepatitis, autoimmune, hemochromatosis...)
* Active neoplastic pathology
* Pregnant or breastfeeding women
* Protected adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2019-04-19 (Actual); Primary Completion 2023-07-19 (Estimated); Study Completion 2024-07-19 (Estimated)

PRIMARY OUTCOMES:
NAFLD and significant fibrosis (≥ F2) | Visit 2
  NAFLD will be defined by the presence of steatosis at ultrasound concomitant with at least one metabolic risk factor among overweight/obesity, type 2 diabetes, dyslipidemia. The severity of NAFLD will be determined by the presence of significant fibrosis (≥F2) by noninvasive measures (either serum markers or transient elastography).

SECONDARY OUTCOMES:
Severity of the coronary lesions | Visit 1
  Based on the results of the coronary angiography, patients will be classified according to the severity of CAD as follows: no CAD, stable CAD (less than 50% stenosis, 1 vessel CAD with > 50% stenosis, 2 vessels CAD with > 50% stenosis, 3 vessels CAD with > 50% stenosis), and acute coronary syndrome.
Correlation between the histological severity of NAFLD and the severity of coronary lesions | 51 months after the start of the study
  The severity of the coronary lesions will be defined as follows : absent, stable coronary lesions (significant >=50% or non significant coronary atheroma), acute coronary syndrome
Analyse of clinical factors associated with the severity of coronary lesions according to the presence or absence of NAFLD | 51 months after the start of the study
  The severity of the coronary lesions will be defined as follows : absent, stable coronary lesions (significant >= 50% or non significant coronary atheroma), acute coronary syndrome
Analyse of the metabolomic signature associated with the severity of coronary lesions according to the presence and severity of NAFLD | Visit 1 and 2
  The severity of the coronary lesions will be defined as follows : absent, stable coronary lesions (significant >=50%or non significant coronary atheroma), acute coronary syndrome

CONTACTS AND LOCATIONS:
Locations (1):
- Pitié Salpêtrière Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No